CLINICAL TRIAL: NCT04356508
Title: COVID-19: A Pilot Study of Adaptive Immunity and Anti-PD1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr Gerry Gin Wai Kwok (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Dr Gerry Gin Wai Kwok, Doctor, Queen Mary Hospital, Hong Kong
Organization: Queen Mary Hospital, Hong Kong (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW20213
Record Dates: First submitted 2020-04-10; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; SARS-CoV-2; 2019-nCoV; Pneumonia, Viral
Keywords: COVID-19; SARS-CoV-2; 2019-nCoV; Coronavirus; Anti-PD1; Nivolumab
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Coronavirus Infections | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (n=10) (Experimental): Nivolumab + best supportive care
  Interventions: Drug: Nivolumab
- Non-intervention (n=5) (No Intervention): Best supportive care

INTERVENTIONS:
Drug: Nivolumab — Single dose at 0.3mg/kg
  Other Names: Opdivo
  Arms: Intervention (n=10)

SUMMARY:
This is an open-label, controlled, single-centre pilot study of nivolumab in adult patients with COVID-19. This clinical study aims to evaluate efficacy of anti-PD1 antibody in relation to viral clearance and its safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 by RT-PCR for SARS-CoV-2
* Clinically stable with disease severity defined as mild or moderate (mild disease is defined as symptoms with or without lung infiltrates on chest X-Ray or CT imaging; moderate disease is defined as lung infiltrates with evidence of type 1 respiratory failure)
* Asymptomatic patients may be enrolled if patients have obvious radiographic changes on chest or CT radiography deemed to be related to COVID-19

Exclusion Criteria:

* Active cancer, rheumatological and autoimmune conditions
* Transplant recipients, or patients on active immunosuppressants
* Chronic organ impairment, or documented or suspected concomitant infections (including chronic viral hepatitis B and hepatitis C) other than SARS-CoV-2
* Lactating mothers and women who are pregnant or intending to become pregnant
* Acute respiratory distress syndrome, evidence of myocardial injury, disseminated intravascular coagulopathy, organ failure, hemophagocytosis, shock, respiratory distress, or need for mechanical ventilation, AICU admission, or high flow oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-04-14 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Viral clearance kinetics | From diagnosis to recovery, assessed up to 6 months
  Viral load changes in NPS based on SARS-CoV-2 RT-PCR

SECONDARY OUTCOMES:
Treatment-related adverse events of nivolumab (Intervention arm only) | Up to 1 year after nivolumab dosing
  Incidence and severity of treatment-related adverse events
Lymphocyte kinetics | On days 1, 4, 6, 8, 10 and 28 from study enrollment
  Changes in lymphocyte counts
Cytokine kinetics | On days 1, 4, 6, 8 and 10 from study enrollment
  Changes in cytokine levels (e.g. IL-1B, IL-2, IL-6, TNFa)
Length of inpatient stay due to COVID-19 | From hospital admission to discharge, assessed up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerry Gin Wai Kwok, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong